CLINICAL TRIAL: NCT02559414
Title: Antiplatelet Therapy in HIV - Antiplatelet and Immune Modulating Effects of Aspirin or Clopidogrel in Subjects With HIV
Brief Title: Antiplatelet Therapy in HIV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 14-02104
Record Dates: First submitted 2015-03-10; First posted 2015-09-24 (Estimated); Results first posted 2017-09-11 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-09

CONDITIONS: HIV; Cardiovascular Diseases; Inflammation
MeSH Terms: conditions — Cardiovascular Diseases; Inflammation | interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): This arm of 10 subjects will be assigned randomly via a computer generated treatment sequence, and then be given no antiplatelet medication.
- Aspirin (Active Comparator): This arm of 20 subjects will be assigned randomly via a computer generated treatment sequence, and then be given aspirin.
  Interventions: Drug: Aspirin
- Clopidogrel (Active Comparator): This arm of 20 subjects will be assigned randomly via a computer generated treatment sequence, and then be given clopidogrel.
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Aspirin
  Arms: Aspirin
Drug: Clopidogrel
  Arms: Clopidogrel

SUMMARY:
The proposed study will add to the growing understanding of platelet activity and platelet inhibition in subjects with HIV. It will examine the relationship between platelet activity and its inhibition by antiplatelet therapy (aspirin monotherapy and clopidogrel monotherapy) in this high-risk cohort. Furthermore, it will provide important data on the mechanism of platelet activity and its inhibition using biomarkers of platelet activity, inflammation, immune activity and endothelial function and genetic expression profiling.

DETAILED DESCRIPTION:
There is substantial evidence that the risk of serious non-AIDS conditions, such as cardiovascular disease, kidney disease, liver disease, and non-AIDS-defining malignancies, is increased in persons with HIV infection as compared to the general population. HIV-induced activation of inflammatory and coagulation pathways have been implicated in this increased risk. However, causative mechanisms linking HIV, inflammation, and increased risk of non-AIDS diseases are poorly described. The investigators are interested in studying the link between HIV induced inflammation and cardiovascular disease. Inflammation mediates many aspects of disease pathogenesis in atherosclerosis, involving diverse cell types and mediating signals. Specifically, platelets have been implicated in atherosclerosis because of their pro-inflammatory and thrombogenic effects. Moreover, clinical studies have demonstrated the importance of platelet activity in coronary artery atherosclerosis and thrombosis. Whereas there is a great understanding of the pathogenesis of cardiac disease, there is a wide knowledge gap in the understanding of mechanisms of cardiovascular disease in patients with HIV.

A recent study by the investigators demonstrated that platelet activity is heightened in subjects with HIV. Following 1-week of low-dose aspirin, platelet activity was inhibited. A surprising finding of this study demonstrated that antiplatelet therapy with 1 week of aspirin (325mg dose x1 day followed by 81mg daily) improved immune activity in subjects with HIV. The current study is being performed to replicate those findings when compared with a control group. Moreover, it remains unknown if the finding was specific to aspirin or whether the results were attributed to the antiplatelet effect of the drug. Clopidogrel is another antiplatelet therapy that targets the P2Y12 receptor (a different mechanism than aspirin) that has been shown to lower the risk of cardiovascular events in various clinical settings. The doses of aspirin and clopidogrel the investigators will be employing have been tested in hundreds of studies with well-known benefits and risks. The investigators believe that understanding the mechanistic role of platelet inhibitors in the setting of HIV will help uncover a new strategic pathway of HIV pathogenesis. Also, subjects with HIV are at increased risk for cardiovascular events and understanding the platelet inhibition of aspirin and clopidogrel will help establish better designs for future trials aimed at preventing these events in HIV infected persons.

The investigators have demonstrated that platelet activation is increased in HIV infection and can be attenuated by low-dose aspirin in a non-randomized study without a control group. Therefore, the Specific Aims of the study to be established are as follows:

* The effect of aspirin versus control on markers of platelet activity, inflammation, immune activity, and endothelial function.
* The effect of Clopidogrel versus control on markers of platelet activity, inflammation, immune activity, and endothelial function.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection
* Current Antiretroviral Therapy with no change in regimen in the 12 weeks prior to study entry and no plans to change ART for the study duration
* Ability to sign consent and comply with the protocol

Exclusion Criteria:

* Known CD4+ T cell counts < 200 cells/mm3 during the 6 months prior to study entry
* Established cardiovascular disease (thereby necessitating antiplatelet therapy)
* NSAID use in the past week (including aspirin)
* Unable to be off NSAIDs for the duration of the trial
* Any antiplatelet or antithrombotic use
* Allergy to aspirin or clopidogrel
* Pregnancy
* Chronic kidney disease (GFR<45 ml/min)
* AIDS
* Active drug or alcohol use that would interfere with adherence to study requirements
* Any known bleeding disorder
* Use of regularly prescribed medication such as steroids, or immunosuppressive agents
* Known anemia (Hb <8mg/dL)
* Thrombocytopenia (platelet count <75) or thrombocytosis (Platelet count >600)

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S Berger, MD, Principal Investigator — NYU School of Medicine
Locations (2):
- United States (2):
  - Bellevue Hospital, New York, New York
  - NYU Langone Medical Center, New York, New York

REFERENCES:
- [Background] Berger JS, Lala A, Krantz MJ, Baker GS, Hiatt WR. Aspirin for the prevention of cardiovascular events in patients without clinical cardiovascular disease: a meta-analysis of randomized trials. Am Heart J. 2011 Jul;162(1):115-24.e2. doi: 10.1016/j.ahj.2011.04.006. PMID 21742097
- [Background] Berger JS, Roncaglioni MC, Avanzini F, Pangrazzi I, Tognoni G, Brown DL. Aspirin for the primary prevention of cardiovascular events in women and men: a sex-specific meta-analysis of randomized controlled trials. JAMA. 2006 Jan 18;295(3):306-13. doi: 10.1001/jama.295.3.306. PMID 16418466
- [Background] CAPRIE Steering Committee. A randomised, blinded, trial of clopidogrel versus aspirin in patients at risk of ischaemic events (CAPRIE). CAPRIE Steering Committee. Lancet. 1996 Nov 16;348(9038):1329-39. doi: 10.1016/s0140-6736(96)09457-3. PMID 8918275
- [Background] Solomon Tsegaye T, Gnirss K, Rahe-Meyer N, Kiene M, Kramer-Kuhl A, Behrens G, Munch J, Pohlmann S. Platelet activation suppresses HIV-1 infection of T cells. Retrovirology. 2013 May 1;10:48. doi: 10.1186/1742-4690-10-48. PMID 23634812
- [Derived] Marcantoni E, Garshick MS, Schwartz T, Ratnapala N, Cambria M, Dann R, O'Brien M, Heguy A, Berger JS. Antiplatelet Effects of Clopidogrel Vs Aspirin in Virologically Controlled HIV: A Randomized Controlled Trial. JACC Basic Transl Sci. 2022 Oct 5;7(11):1086-1097. doi: 10.1016/j.jacbts.2022.06.002. eCollection 2022 Nov. PMID 36687270

RESULTS

PARTICIPANT FLOW:
Groups:
- Aspirin: This arm of 20 subjects will be assigned randomly via a computer generated treatment sequence, and then be given aspirin.
  Aspirin
- Clopidogrel: This arm of 20 subjects will be assigned randomly via a computer generated treatment sequence, and then be given clopidogrel.
  Clopidogrel
Period: Overall Study
Arm/Group | Control | Aspirin | Clopidogrel
Started | 11 | 22 | 22
Completed | 10 | 20 | 20
Not Completed | 1 | 2 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Other | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Aspirin | Clopidogrel | Total
Number analyzed (Participants) | 11 | 22 | 22 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 20 | 19 | 50
  >=65 years | 0 | 2 | 3 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 10 | 23
  Male | 5 | 15 | 12 | 32

OUTCOME MEASURES:

1. Primary Outcome: Percentage Platelet Aggregation in PRP After Stimulation With Arachidonic Acid 1600 μM for 5 Min
Description: The primary objective of these analyses will be to compare the effects of aspirin versus control and clopidogrel versus control for the outcome of platelet activity. Aspirin is expected to decrease arachidonic acid-induced platelet aggregation by 50% versus control. Clopidogrel is expected to decrease ADP-induced platelet aggregation by 50% versus control.
Time Frame: Baseline, 14 Days
Measure: Mean (Standard Error); unit: %aggregation
Groups:
- Placebo Baseline: This arm of 10 subjects will be assigned randomly via a computer generated treatment sequence, and then be given no antiplatelet medication.
Arm/Group | Placebo Baseline | Placebo Follow up | Aspirin Baseline | Aspirin Randomization | Clopidogrel Baseline | Clopidogrel Randomization
Number analyzed (Participants) | 10 | 9 | 14 | 13 | 21 | 16
%aggregation | 72.35 (5.71) | 79.11 (3.15) | 72.79 (5.11) | 26.77 (7.61) | 71.07 (6.16) | 65.00 (8.16)

2. Secondary Outcome: Percentage Platelet Aggregation in PRP After Stimulation With ADP 5μM for 5 Min
Time Frame: Baseline, 14 Days
Measure: Mean (Standard Error); unit: %aggregation
Arm/Group | Placebo Baseline | Placebo Follow up | Aspirin Baseline | Aspirin Randomization | Clopidogrel Baseline | Clopidogrel Randomization
Number analyzed (Participants) | 10 | 9 | 14 | 13 | 21 | 16
%aggregation | 69.45 (9.04) | 80.33 (2.77) | 82.04 (2.44) | 62.00 (5.50) | 78.86 (3.45) | 39.88 (7.95)

3. Secondary Outcome: Percentage Monocyte-Platelet Aggregates
Description: Secondary objectives will compare the effect of each antiplatelet therapy drug on biomarkers related to inflammation
Time Frame: 14 Days
Measure: Mean (Standard Error); unit: %aggregation
Arm/Group | Placebo Baseline | Placebo Follow up | Aspirin Baseline | Aspirin Randomization | Clopidogrel Baseline | Clopidogrel Randomization
Number analyzed (Participants) | 10 | 9 | 14 | 13 | 21 | 16
%aggregation | 69.45 (9.04) | 80.33 (2.77) | 82.04 (2.44) | 62.00 (5.50) | 78.86 (3.45) | 39.88 (7.95)

4. Secondary Outcome: Percentage Monocyte-Platelet Aggregates
Description: Secondary objectives will compare the effect of each antiplatelet therapy drug on biomarkers related to immune activity
Time Frame: 14 Days
Measure: Mean (Standard Error); unit: %aggregation
Arm/Group | Placebo Baseline | Placebo Follow up | Aspirin Baseline | Aspirin Follow up | Clopidogrel Baseline | Clopidogrel Follow up
Number analyzed (Participants) | 8 | 7 | 10 | 8 | 16 | 13
%aggregation | 15.53 (1.28) | 15.43 (2.07) | 13.15 (1.15) | 14.96 (1.33) | 16.03 (1.47) | 14.85 (0.85)

5. Secondary Outcome: Percentage Leukocyte-Platelet Aggregate
Description: Secondary objectives will compare the effect of each antiplatelet therapy drug on biomarkers related to endothelial function.
Time Frame: 14 Days
Measure: Mean (Standard Error); unit: %aggregation
Arm/Group | Placebo Baseline | Placebo Follow up | Aspirin Baseline | Aspirin Randomization | Clopidogrel Baseline | Clopidogrel Randomization
Number analyzed (Participants) | 8 | 7 | 15 | 11 | 17 | 14
%aggregation | 14.06 (1.24) | 13.84 (1.97) | 11.18 (0.90) | 12.11 (1.01) | 13.06 (0.83) | 12.29 (0.88)

ADVERSE EVENTS:
Arm/Group | Placebo Baseline | Placebo Follow up | Aspirin Baseline | Aspirin Randomization | Clopidogrel Baseline | Clopidogrel Randomization
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9 | 0/14 | 0/13 | 0/21 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/9 | 0/14 | 0/13 | 0/21 | 0/16
Other Adverse Events (participants affected / at risk) | 1/10 | 0/9 | 0/14 | 0/13 | 0/21 | 0/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Baseline (N=10) | Placebo Follow up (N=9) | Aspirin Baseline (N=14) | Aspirin Randomization (N=13) | Clopidogrel Baseline (N=21) | Clopidogrel Randomization (N=16)
Diverticulitis with mesenteric thrombophlebitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — The subject's symptoms occurred after enrollment, but well before study drug administration.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Baseline (N=10) | Placebo Follow up (N=9) | Aspirin Baseline (N=14) | Aspirin Randomization (N=13) | Clopidogrel Baseline (N=21) | Clopidogrel Randomization (N=16)
stomach irritation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No